CLINICAL TRIAL: NCT01813448
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Dose Escalation Study to Assess the Safety, Tolerability and Pharmacokinetics of Single and Multiple Ascending Doses of Fidaxomicin in Healthy Male Japanese and Caucasian Subjects
Brief Title: A Study to Assess the Safety, Tolerability and Pharmacokinetics of Single and Multiple Ascending Doses of Fidaxomicin in Healthy Male Japanese and Caucasian Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 2819-CL-3001
Record Dates: First submitted 2013-03-15; First posted 2013-03-19 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Pharmacokinetics of Fidaxomicin; Healthy Subjects
Keywords: Fidaxomicin; OPT-80; Healthy Subjects
MeSH Terms: interventions — Fidaxomicin; OPT 80

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort 1: Fidaxomicin low dose in Japanese males (Experimental)
  Interventions: Drug: Fidaxomicin
- Cohort 2: Fidaxomicin high dose in Japanese males (Experimental)
  Interventions: Drug: Fidaxomicin
- Cohort 3: Fidaxomicin high dose in Caucasian males (Experimental)
  Interventions: Drug: Fidaxomicin
- Matching Placebo in Caucasian males (Placebo Comparator)
  Interventions: Drug: Placebo
- Matching Placebo in Japanese males (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fidaxomicin — oral
  Other Names: OPT-80; Dificlir; Dificid
  Arms: Cohort 1: Fidaxomicin low dose in Japanese males; Cohort 2: Fidaxomicin high dose in Japanese males; Cohort 3: Fidaxomicin high dose in Caucasian males
Drug: Placebo — oral
  Arms: Matching Placebo in Caucasian males; Matching Placebo in Japanese males

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics (PK) of single and multiple ascending doses of fidaxomicin in healthy subjects. This study will also compare the safety, tolerability and PK of single and multiple doses of fidaxomicin in healthy Japanese and Caucasian subjects.

DETAILED DESCRIPTION:
Eligible subjects will check into the unit on Day-2 and remain confined to the clinical unit until Day 17.

Cohorts 2 and 3, which may run in parallel, will only be enrolled after review of the available safety data of Cohort 1 by the Safety Review Team.

ELIGIBILITY:
Inclusion Criteria:

1. Male subject and their female spouse/partners who are of childbearing potential must be using highly effective contraception consisting of two forms of birth control (one of which must be a barrier method) starting at Screening and continuing throughout the study period and for 90 days after final study drug administration
2. Male subject must not donate sperm starting at Screening and throughout the study period and for at least 90 days after final study drug administration

   Inclusion Criteria for Japanese Subjects
3. The subject is a healthy Japanese male who maintains the Japanese lifestyle, including diet and has a body mass index (BMI) of 18.0 to 28.0 kg/m2, inclusive.

   Inclusion Criteria for Caucasian Subjects
4. The subject is a healthy Caucasian male and has a BMI of 18.0 to 32.0 kg/m2, inclusive

Exclusion Criteria:

1. The subject has any clinically significant disease history
2. The subject has a history of or current C.difficile infection or history of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (history of appendectomy, hernia repair, and/or cholecystectomy is permitted)
3. The subject has any clinically significant abnormality
4. The subject has a resting (i.e., seated for 5 minutes) pulse <40 or >90 beats per minute (bpm) at Screening or Day -2
5. The subject has hypertension (defined as seated systolic blood pressure [SBP] >140 mmHg or seated diastolic blood pressure [DBP] >90 mmHg) or hypotension (defined as seated SBP <90 mmHg or seated DBP <50 mmHg) at Screening or Day -2
6. The subject has/had a symptomatic, viral, bacterial (including upper respiratory infection), or fungal (non-cutaneous) infection within 1 week prior to clinic check-in on Day -2
7. The subject has a history of chronic diarrhea or constipation
8. The subject has a positive result for hepatitis C antibodies or hepatitis B surface antigen at Screening or has a known positive history of human immunodeficiency virus (HIV)
9. The subject has a known or suspected allergy or hypersensitivity to any of the components of fidaxomicin, the macrolide antibacterial class of compounds, or a history of multiple and/or severe allergies to drugs or foods or a history of severe anaphylactic reactions

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2013-02; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) of fidaxomicin in plasma (single dose): Lag time (tlag) | Days 1-5 (14 times)
PK of fidaxomicin plasma (single dose): Time to attain maximum concentration (tmax) | Days 1-5 (14 times)
PK of fidaxomicin in plasma (single dose): Maximum Concentration (Cmax) | Days 1-5 (14 times)
PK of fidaxomicin in plasma (single dose): Area Under the Plasma Concentration - Time Curve (AUC) from Time Zero to Time of Last Measurable Concentration (AUClast) | Days 1-5 (14 times)
PK of fidaxomicin in plasma (single dose): AUC - Time Curve from Time Zero to Infinity (aucinf) | Days 1-5 (14 times)
PK of fidaxomicin in plasma (single dose): AUC - Time Curve from Time Zero to 12 hours (AUC 0-12h) | Days 1-5 (14 times)
PK of fidaxomicin in plasma (single dose): Total Body Clearance after Single Dose (CL/F) | Days 1-5 (14 times)
PK of fidaxomicin in plasma (single dose): Apparent Volume of Distribution During Terminal Phase (Vz/F) | Days 1-5 (14 times)
PK of fidaxomicin in plasma (last dose): Apparent Volume of Distribution During Terminal Phase (Vz/F) | Days 15-17 (11 times)
PK of fidaxomicin in plasma (single dose): Apparent Terminal elimination Half-life (t 1/2) | Days 1-5 (14 times)
  Single Dose
PK of fidaxomicin in plasma (last dose): Apparent Terminal elimination Half-life (t 1/2) | Days 15-17 (11 times)
  Single Dose
PK of fidaxomicin in plasma (single dose): Trough levels | Days 6, 7, 10, and 12 (pre-morning dose)
PK of fidaxomicin in plasma (last dose): tmax at Steady State (tmax, ss) | Days 15-17 (11 times)
  Last Dose
PK of fidaxomicin in plasma (last dose): Cmax at Steady State (Cmax, ss) | Days 15-17 (11 times)
  Last Dose
PK of fidaxomicin in plasma (last dose): AUC Over the dosing Interval (AUCtau) | Days 15-17 (11 times)
PK of fidaxomicin in plasma (last dose): CL/F at Steady State (CL/F ss) | Days 15-17 (11 times)
PK of fidaxomicin in plasma (last dose): Peak: Trough Ratio (PTR) | Days 15-17 (11 times)
PK of fidaxomicin in plasma (last dose): Accumulation Ratio (Racc) | Days 15-17 (11 times)
PK of fidaxomicin in plasma (last dose): Pre-dose Plasma Concentration Determined Directly from the Concentration-Time Profile (Ctrough) | Days 15-17 (11 times)
PK of fidaxomicin in urine (last dose): Cumulative Amount of Drug Excreted in the urine from Time Zero to Time of Last Measurable Concentration (Aelast) | Days 1-5 (6 times)
PK of fidaxomicin in urine (single dose): Percent Fraction of Administered Drug Excreted Unchanged in the urine from Time Zero to Time of Last Measurable Concentration (% Aelast ) | Days 1-5 (6 times)
PK of fidaxomicin in urine (single dose): Cumulative Amount of Drug Excreted in the Urine from time Zero to Infinity after Single Dose (Aeinf) | Days 1-5 (6 times)
PK of fidaxomicin in urine (single dose): Percent Fraction of administered drug excreted unchanged in the urine from time Zero to Infinity after Single Dose (% Aeinf) | Days 1-5 (6 times)
PK of fidaxomicin in urine (single dose): Renal Clearance (CL/R | Days 1-5 (6 times)
PK of fidaxomicin in urine (last dose): Cumulative Amount of Drug Excreted in the urine over the dosing Interval at Steady State (Aetau) | Day 15 (1 time)
PK of fidaxomicin in urine (last dose): Percent Fraction of Administered Drug Excreted Unchanged in the Urine over the Dosing Interval at Steady State (% Aetau) | Day 15 (1 time)
PK of fidaxomicin in urine (last dose): Renal Clearance at Steady State (CLR,ss) | Day 15 ( 1 time)
PK of fidaxomicin in feces (single dose): Amount of Drug Excreted in the Feces (Ae) | Days 1-5 (5 times)
PK of fidaxomicin in feces (last dose): Amount of Drug Excreted in the Feces (Ae) | Days 15-17 (first bowel movement (BM) following the last dose to be collected)
PK of fidaxomicin in feces (single dose): Percent Fraction of Administered Drug Excreted Unchanged in the Feces (%Ae) | Days 1-5 (5 times)
PK of fidaxomicin in feces (last dose): Percent Fraction of Administered Drug Excreted Unchanged in the Feces (%Ae) | Days 15-17 (first BM following the last dose to be collected)

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (1):
- Parexel, Glendale, California, United States